CLINICAL TRIAL: NCT04177732
Title: Assessment of Efficacy of Calprotectin and Cross-linked N-telopeptides of Type I Collagen Levels in Crevicular Fluid as a Biomarker in Patients With Peri-implantitis: A Clinical Study
Brief Title: Assessment of Efficacy of Calprotectin and Cross-linked N-telopeptides
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Mansour Assery (Other)
Responsible Party: Sponsor-Investigator, Mansour Assery, Consultant in Prosthodontics & Dental Implant, Riyadh Elm University
Organization: Riyadh Elm University (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: Calprotectin-N-telopeptides
Record Dates: First submitted 2019-11-22; First posted 2019-11-26 (Actual); Last update posted 2019-12-02 (Actual); Status verified 2019-11

CONDITIONS: Peri-Implantitis; Dental Implant Failed
Keywords: biomarkers; Calprotectin; Cross-linked N-telopeptides
MeSH Terms: conditions — Peri-Implantitis

STUDY DESIGN:
Intervention Model Description: Group A: Healthy peri-implant status Group B: Presence of peri-implant diseases
Masking Description: No masking
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Healthy peri-implant status (Other): Patient with healthy peri-implant status
  Interventions: Diagnostic Test: Collection of sulcular (crevicular) fluid; Diagnostic Test: Probing depth; Diagnostic Test: Bleeding on probing; Diagnostic Test: Gingival index; Diagnostic Test: Bone loss rate of alveolar bone
- Presence of peri-implant diseases (Other): Patients with presence of peri-implant diseases
  Interventions: Diagnostic Test: Collection of sulcular (crevicular) fluid; Diagnostic Test: Probing depth; Diagnostic Test: Bleeding on probing; Diagnostic Test: Gingival index; Diagnostic Test: Bone loss rate of alveolar bone

INTERVENTIONS:
Diagnostic Test: Collection of sulcular (crevicular) fluid — Sterile paper strips will be used for collecting crevicular fluid
Diagnostic Test: Probing depth — Williams SE manual probe will be used to measure the probing depth
Diagnostic Test: Bleeding on probing — Williams SE manual probe will be used to probe the sulcus a oserve the gingival reaction
Diagnostic Test: Gingival index — Modified Löe and Silness criteria will be used for evaluating the gingival index score
Diagnostic Test: Bone loss rate of alveolar bone — Using modification of criteria described by Schei et al, bone loss rate of alveolar bone will be analyzed on radiographic assessment

SUMMARY:
The study aims to assess the efficacy of Calprotectin and cross-linked N-telopeptides of type I collagen levels in crevicular fluid as a biomarker in patients with peri-implantitis.

DETAILED DESCRIPTION:
Ethical approval will be obtained from the ethical committee of the Riyadh Elm University and written consent will be obtained from all the patients after explaining in detail the entire research protocol.

Inclusion criteria for the present study:

* 10 patients who underwent dental implant procedure five to ten years ago; among these- 5 patients will be with healthy peri-implant status and 5 patients with presence of peri-implant diseases
* Patients of comparable age and gender distribution- Patients within the age group of 25 to 45 years; and 3 males and 2 females in peri-implant diseases group and 3 males and 2 females in healthy peri-implant status group
* Patients with negative history of any systemic illness, metabolic disease.
* Patients with negative history of antibiotic therapy in past ninety days.

After collecting the PICF and GCF, examination of probing depth (PD), bleeding on probing (BOP) and gingival index (GI) will be done.Modified Löe and Silness criteria will be used for evaluating the GI score.Using modification of criteria described by Schei et al, bone loss rate of alveolar bone will be analyzed on radiographic assessment. Periodontal sites with PD of equal to or more than 3mm with GI score of equal to or more than 1mm and presence or absence of BOP, will be categorized as peri-implant disease sites. Periodontal sites with PD of less than 3mm with GI score of 0 and absence of BOP will be categorized as healthy implant sites. Sterile paper strips will be used for collecting PICF samples, followed by PICF sample preparation using modified criteria described previously in the literature. Isolation of the PICF sampling sites will be done using cotton roles. This will be followed by removal of supra-gingival plaques and gentle air drying. Insertion of the periopaper will be done into the peri-implant crevice and will be kept there for thirty seconds. Periotron will be used for measuring the volume of PICF. Further, all the samples will be sent to laboratory where ELISA technique will be used for measuring the calprotectin

ELIGIBILITY:
Inclusion Criteria:

Exclusion Criteria:

* Patients with history of any systemic illness, metabolic disease.
* Patients with history of antibiotic therapy in past ninety days.

Ages: 25 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 10 (Estimated)
Dates: Start 2019-12-10 (Estimated); Primary Completion 2020-02-01 (Estimated); Study Completion 2020-04-01 (Estimated)

PRIMARY OUTCOMES:
Calprotectin concentration in GCF | 3 weeks
  One of inflammation biomarkers found in gingival crevicular fluid (GCF) that are associated with bone inflammation
Cross-linked N-telopeptides concentration in GCF | 3 weeks
  One of inflammation biomarkers found in gingival crevicular fluid (GCF) that are associated with bone inflammation

IPD SHARING:
Plan to Share IPD: Undecided